CLINICAL TRIAL: NCT01750385
Title: Bacteremia and Procalcitonin Levels in Peroral Endoscopic Myotomy for Achalasia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: B2012-089
Record Dates: First submitted 2012-11-20; First posted 2012-12-17 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Esophageal Achalasia
Keywords: Esophageal Achalasia; antibiotic prophylaxis; blood culture; procalcitonin levels
MeSH Terms: conditions — Esophageal Achalasia | interventions — Second Generation Cephalosporins

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- no antibiotic prophylaxis (Active Comparator): These patients are in no antibiotic prophylaxis group will not be administered antibiotic prophylactically.
  Interventions: Drug: no antibiotic prophylaxis
- second-generation cephalosporin (Active Comparator): These patients are in antibiotic prophylaxis group will be administered second-generation cephalosporin prophylactically.
  Interventions: Drug: second-generation cephalosporin

INTERVENTIONS:
Drug: no antibiotic prophylaxis — These patients are in no antibiotic prophylaxis group will not be administered antibiotic prophylactically.
  Arms: no antibiotic prophylaxis
Drug: second-generation cephalosporin — These patients are in antibiotic prophylaxis group will be administered second-generation cephalosporin prophylactically.
  Arms: second-generation cephalosporin

SUMMARY:
Peroral Endoscopic Myotomy (POEM) is a novel, promising endoscopic technique for achalasia because it is safer and more effective than traditional Heller's myotomy. However, the issue of antibiotic prophylaxis in POEM has evoked considerable controversy recently. Therefore, we conduct this study to elucidate the status of POEM-related bacteremia and procalcitonin levels in order to preliminary observe whether antibiotic prophylaxis is needed.

DETAILED DESCRIPTION:
Objective: To elucidate the status of POEM-related bacteremia and procalcitonin levels in order to preliminary observe whether antibiotic prophylaxis is needed.

Interventions: Patients with achalasia diagnosed by symptoms, endoscopy and barium swallow eligible for POEM are randomized to either use antibiotic prophylactically or not.

Main outcome measurements: Blood culture positive incidence; secondary outcomes are procalcitonin levels, C-reactive protein levels, white blood cell counts and so on.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of esophageal achalasia
* Ready to have the treatment as POEM and no contraindication of POEM
* Ability to get informed consent

Exclusion Criteria:

* Patients who had indications for antibiotic prophylaxis as determined by the American Society for Gastrointestinal Endoscopy
* Patients who had received antibiotics for any reason within the previous 7days
* Patients who had possible signs of any infection at the time of the procedure
* Patients who had chronic inflammatory diseases need hormonotherapy : such as rheumatic arthritis or inflammatory bowel diseases.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-04 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Blood culture positive incidence | after 12 hours of POEM
  To compare the positive incidence of blood cultures between antibiotic prophylaxis and no antibiotic prophylaxis.

SECONDARY OUTCOMES:
procalcitonin level | after 12 hours of POEM
  To observe the changes of procalcitonin levels after POEM in which no antibiotic is administered.
  To compare the procalcitonin levels between antibiotic prophylaxis and no antibiotic prophylaxis.

OTHER OUTCOMES:
clinical manifestation | during hospital stay and up to 1 week
  To observe the changes of temperature, heart rate, respiratory rate, white blood cell counts, neutrophile granulocyte counts in perioperative period.

CONTACTS AND LOCATIONS:
Overall Officials: Ping-Hong Zhou, M.D,PhD, Study Director — Fudan University